CLINICAL TRIAL: NCT01269476
Title: Phase 1 Safety and Pharmacokinetics of Methane Sulfonylfluoride (MSF or SNX-001) After Single and Multiple Oral Dose Administration in Healthy Adult Aged Volunteers
Brief Title: Safety and Pharmacokinetics of SNX-001 in Healthy Aged Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SeneXta Therapeutics SA (Industry)
Responsible Party: Dr. Enrico Braglia, SeneXta Therapeutics SA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNX-001-PH1-09; 2009-011335-13 (EudraCT Number)
Record Dates: First submitted 2010-09-22; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Safety
MeSH Terms: interventions — methanesulfonyl fluoride; Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SNX-001 (Experimental)
  Interventions: Drug: SNX-001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNX-001 — 3.6, 7.2, or 10.8 mg single dose or t.i.w.
  Other Names: methanesulfonyl fluoride; MSF
  Arms: SNX-001
Drug: Placebo — Same volumes and frequency as active.
  Other Names: Oil vehicle
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, group-sequential, placebo-controlled, safety and pharmacokinetic study in healthy, aged volunteers.

Objectives:

1. to confirm the previously reported safety profile of oral SNX-001 after single and multiple doses of 3.6, 7.2 or 10.8 mg compared to placebo
2. to establish SNX-001 pharmacokinetic profile.

DETAILED DESCRIPTION:
This study is an exploratory study designed as a group sequential single and multiple escalating dose, double-blind within cohort, randomized, placebo controlled study to investigate the safety and tolerability as well as the pharmacokinetics and pharmacodynamics of SNX-001 given as oral doses in aged volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females
* Physically and mentally healthy subjects
* Body weight >60 kg and body weight ≤ 100 kg

Exclusion Criteria:

* Evidence of any clinically significant hepatic, renal, gastrointestinal, cardiovascular, pulmonary, haematological, psychiatric, neurological or other significant acute or chronic abnormalities
* History of general malignant diseases
* Evidence of myasthenic weakness
* Acute infection or any other febrile illness

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Relationship of clinical safety measurements to dose | Throughout 14-day study period (Days 1, 2, 3, 10, 12, 13, 14) and 7 days after last dose (Day 21)
  Adverse events (AEs), vital signs, electrocardiogram (ECG), Acetylcholinesterase (AChE) inhibition, laboratory parameters after single and multiple dose administration

SECONDARY OUTCOMES:
Effect of dose on pharmacokinetic (PK) parameters | After single (Day 1) and multiple (Day 12) doses
  Pharmacokinetic parameters after single and multiple dose administration of SNX-001 (3.6, 7.2 and 10.8 mg)

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Sahlmann, MD, Principal Investigator — Scope Life Sciences GmbH
Locations (1):
- Scope Life Sciences GmbH, Hamburg, Germany